CLINICAL TRIAL: NCT05990686
Title: Preemptive Intravenous Paracetamol Plus Tramadol Versus Preemptive Intravenous Fentanyl in Day Case Surgeries
Brief Title: Paracetamol Plus Tramadol Versus Fentanyl in Day Case Surgeries
Status: Recruiting | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Michael Adel Shaker, lecturer of anesthesia and intensive care, Zagazig University
Other Study IDs: 9702/19-10-2022
Record Dates: First submitted 2023-07-29; First posted 2023-08-14 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Tramadol; Fentanyl

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- paracetamol plus tramadol: randomized selection of 66 adult patients
  Interventions: Drug: Tramadol Hydrochloride
- fentanyl: randomized selection of 66 adult patients
  Interventions: Drug: Fentanyl injection

INTERVENTIONS:
Drug: Tramadol Hydrochloride — After routine pre-operative evaluation, standard monitors will be connected to the patients: pulse oximetery, noninvasive blood pressure and electrocardiogram and baseline parameter will be recorded (heart rate, mean arterial pressure and peripheral oxygen saturation). Intravenous (IV) line will be inserted for all patients, and IV fluid will be started.
  Intravenous infusion of 15mg/kg paracetamol together with 1mg/kg tramadol will be started and to be finished before starting of induction of anaesthesia (induction agent will be Propofol 2mg/kg)
  Other Names: tramadol
  Groups: paracetamol plus tramadol
Drug: Fentanyl injection — After routine pre-operative evaluation, standard monitors will be connected to the patients: pulse oximetery, noninvasive blood pressure and electrocardiogram and baseline parameter will be recorded (heart rate, mean arterial pressure and peripheral oxygen saturation). Intravenous (IV) line will be inserted for all patients, and IV fluid will be started...Intravenous injection of 1microgram/kg fentanyl will be given to the patient followed by induction agents ( propofol 2mg/kg).
  .
  Other Names: fentanyl
  Groups: fentanyl

SUMMARY:
Postoperative pain is an important problem, especially for day case surgeries. It has negative effects on patient's hemodynamics and can cause delayed ambulation resulting in prolonged duration of hospital stay and poor patient satisfaction.

Multiple analgesic strategies have been proposed including NSAID, opioids, epidural analgesia. Each of them has its limitations.

In this study the investigators will compare between the effect of preemptive use of paracetamol plus tramadol versus preemptive intravenous fentanyl in controlling postoperative pain

DETAILED DESCRIPTION:
After routine pre-operative evaluation, standard monitors will be connected to the patients: pulse oximetery, non invasive blood pressure and electrocardiogram and baseline parameter will be recorded (heart rate, mean arterial pressure and peripheral oxygen saturation). Intravenous (IV) line will be inserted for all patients, and IV fluid will be started.

Patients will be allocated into two equal groups;

Group (T) (n=66):

Intravenous infusion of 15mg/kg paracetamol together with 1mg/kg tramadol will be started and to be finished before starting of induction of anesthesia (induction agent will be Propofol 2mg/kg)

Group ( F ) (n=66):

Intravenous injection of 1microgram/kg fentanyl will be given to the patient followed by induction agents ( Propofol 2mg/kg).

In both groups intraoperative monitoring of heart rate (beat/min) and mean arterial blood pressure (mm gh) will be documented.

Postoperatively:

In the recovery room and in the surgical ward patient's mean blood pressure and heart rate will be measured and recorded at 1, 2, 4, 6, and 12 hours postoperatively. Also the postoperative pain assessment for all patients will be done by an anesthesiologist (independent observer) at 1, 2, 4, 6 and 12 hours after surgery based on visual analog scale (VAS) ( a 10-cm line labeled with "worst pain imaginable" on the right border and "no pain" on the left border). The patient is instructed to make a mark along the line to represent the intensity of pain currently being experienced.

Standard postoperative analgesia consisted of paracetamol 1gm i.v. after 6 hours. A rescue analgesic diclofenac 75mg IV infusion will be applied to patients if their VAS score was ≥ 3 and if paracetamol had been administered less than 6 hours before. Time of first required dose of rescue analgesic and total rescue analgesic consumption over the 24-h study period will be documented.

Rescue antiemetics will be given to any patient complaining of nausea and vomiting, occurrence of other side effects including bradycardia or hypotension will be recorded and managed (hypotension defined as a decrease in mean arterial pressure (MAP) of more than 20% of baseline value and planned to be treated with crystalloid infusion and 5 mg bolus of ephedrine, Bradycardia is considered if the heart rate (HR) went below 50 b/min and planned to be managed with atropine 0.2-0.5 mg). Patient satisfaction and length of postoperative hospital stay will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for day case surgeries.
* Both sex
* Patient's age 21 - 60 years.
* Patients with ASA physical status I, II.
* BMI 25 - 30 kg m-2.

Exclusion Criteria:

* Uncooperative patients and patients with psychological problems.
* Patients with liver or renal impairment..
* Patients with history of allergy to drug used in the study.
* Patients with chronic pain.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: patients scheduled for a day case surgeries
Sampling Method: Probability Sample
Enrollment: 132 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
postoperative analgesia | immediately postoperative (0 hour), 1 hour, 2 hours , 4 hours, 6 hours and 12 hours
  Assess quality of postoperative analgesia in both groups analogue score (VAS) scale where zero means no pain and ten means worst pain

SECONDARY OUTCOMES:
mean arterial Blood pressure | 5 minutes after start of surgery (intraoperative) , immediately after surgery (0 hour) , 1 hour, 2 hours , 4 hours , 6 hours and 12 hours after surgery
  Compare mean arterial blood pressure in (mm hg) between patients in both groups
rescue analgesic | immediately after surgery (0 hour) , 1 hour, 2 hours , 4 hours , 6 hours and 12 hours after surgery
  document the first time for the need of rescue analgesics
side effects | up to twenty four hours after surgery
  document the incidence of side effects including: bradycardia, hypotension, nausea and vomiting
length of hospital stay | up to twenty four hours after surgery
  Compare the length of hospital stay in both groups
Heart Rate | 5 minutes after start of surgery ( intraoperative), immediately after surgery (0 hour) , 1 hour, 2 hours , 4 hours , 6 hours and 12 hours after surgery
  compare the heart rate in rate per minutes (rpm) between patients in both groups

CONTACTS AND LOCATIONS:
Overall Officials: MICHAEL A shaker, lecturer, Principal Investigator — Zagazig University
Locations (1):
- Zagazig University , Fuculty of Medicine, Zagazig, Sharquia, Egypt